CLINICAL TRIAL: NCT01820533
Title: Survey of Smokers Treated in the ED on Ownership and Usage of Cell Phones
Brief Title: Survey of Smokers Treated in the Emergency Department (ED) on Ownership and Usage of Cell Phones
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0907005437-2; 5R01CA141479-04 (NIH)
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Smoking
Keywords: Smoking; Cellular phones; Low income population
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- smokers
  Interventions: Other: Cell Phone Survey

INTERVENTIONS:
Other: Cell Phone Survey — Eight item survey for smokers being treated in the YNHH Emergency Dept. The survey asks about the type of cell phone(s) subjects have, how much they pay for cell service monthly, housing status, and if they receive any benefit that would qualify them for the Lifeline program.

SUMMARY:
To study ownership and use of cell phones in low-income smokers. This may help us better understand the impact of cell phone ownership plans on low income smokers' access to quitlines. Use of quitlines may be impeded by limited access to landline phones and limited airtime minutes on cell phones.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* speak and understand English
* willing and able to give informed consent
* have smoked more than 100 cigarettes lifetime
* are currently a daily or some day smoker

Exclusion Criteria:

* too ill or unable to consent
* not interested in participation
* actively psychotic or mentally ill and unable to give consent
* in police custody
* resides in an extended care facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be current patients in the Yale New Haven Hospital Emergency Department who were previously identified as smokers.
Sampling Method: Non-Probability Sample
Enrollment: 775 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with lifeline wireless phones | baseline
  The proportion of participants who have lifeline wireless phones (AKA "Medicaid phones").
proportion of participants with limited wireless minutes | baseline
  The proportion of participants with limited wireless minutes each month, stratified by insurance.
proportion of participants with unlimited wireless minutes | baseline
  The proportion of participants with unlimited wireless minutes each month, stratified by insurance status.

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Bernstein, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States